CLINICAL TRIAL: NCT01813461
Title: A Phase 1 Open-Label Mass Balance Study to Evaluate the Pharmacokinetics of Isavuconazole After a Single Oral Dose of 14C-Labeled Isavuconazonium Sulfate in Healthy Male Subjects
Brief Title: Study to Evaluate the Pharmacokinetics of 14C-labeled Isavuconazole Following a Single Oral Dose of 14C-labeled Prodrug Isavuconazonium Sulfate (BAL8557) in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0016
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Pharmacokinetics of 14C-labeled Isavuconazole; Healthy Subjects
Keywords: BAL8557; 14C-labeled isavuconazole; 14C-labeled prodrug isavuconazonium sulfate (BAL8557)/([cyano-14C]ASP9766 sulfate)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 14C-labeled prodrug isavuconazonium sulfate (Experimental): single dose
  Interventions: Drug: 14C-labeled prodrug isavuconazonium sulfate

INTERVENTIONS:
Drug: 14C-labeled prodrug isavuconazonium sulfate — oral

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of 14C-labeled isavuconazole and the routes of excretion and the extent of metabolism of 14C-labeled prodrug BAL8557.

DETAILED DESCRIPTION:
Subjects will be admitted to and stay in a clinical research unit for 23 days. On Day 1, they will receive a single oral dose of BAL8557 and throughout the study period the excretion and metabolism of the study drug will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45 kg and a body mass index of 18 to 32 kg/m2, inclusive.
* The subject's 12-lead electrocardiogram (ECG) is normal at Screening and Day -1; or, if abnormal, the abnormality is not clinically significant, including a QT interval corrected for heart rate using Fridericia's formula (QTcF) of 430 msec or less.
* The subject's clinical laboratory test results at Screening and Day 1 are within normal limits or not clinically significant.
* Results for aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be within the normal range.
* The subject is surgically sterile or agrees to using a highly effective method of contraception to prevent pregnancy during the study and for at least 90 days after dosing on Day 1, and the subject agrees to not donate any sperm for at least 90 days after dosing on Day 1.

Exclusion Criteria:

* The subject has any clinically significant disease history or condition that precludes him from participating in the trial.
* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome
* The subject has a history of bowel obstruction, swallowing disorder, severe gastrointestinal disorders, major gastrointestinal surgery, actively bleeding hemorrhoids, or gastric/duodenal ulcers.
* The subject has irregular bowel habits (< 1 bowel movement per day).
* The subject has had nuclear medicine procedures, computed tomography scans, or significant x-rays (other than dental) within the past 12 months, has had significant occupational radiation exposure, or participated in a radio-labeled study within the last 6 months or participated in more than one radio-labeled study within the last 12 months.
* The subject has a positive test for hepatitis B surface antigen or hepatitis C antibodies at Screening or is known to be positive for human immunodeficiency virus (HIV).
* The subject has/had a symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to clinic admission on Day -1.
* The subject has received a vaccination within the last 30 days prior to study drug administration.
* The subject has a known or suspected allergy to any of the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods (as judged by the Investigator), or a history of severe anaphylactic reactions.
* The subject has used tobacco or nicotine containing products in the last 6 months.
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to Day -1, or over-the-counter medication within 1 week prior to Day -1, with the exception of occasional use of acetaminophen up to 2 g/day.
* The subject has participated in any interventional clinical study or has received any investigational agent within 30 days or 5 half-lives, whichever is longer, prior to the initiation of Screening.
* The subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission on Day -1.
* The subject has taken part in strenuous exercise within 3 days prior to dosing on Day 1.
* The subject anticipates an inability to abstain from caffeine or alcohol use for 48 hours prior to clinic admission on Day -1 and throughout the duration of the study; or from grapefruit, grapefruit juice, star fruit, or Seville oranges or any products containing these items from 72 hours prior to clinic admission on Day -1 and throughout the duration of the study.
* The subject has a recent history (within the last 2 years) of drug or alcohol abuse or a positive drug screen.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Radioactivity in whole blood and in plasma: Area under the concentration-time curve (AUC) from time of dosing to infinity (AUCinf) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 312, 360, 408, 456, and 504 hours after radioactive dose. If subjects are not discharged on Day 22, blood will be collected at 576 and 648 hours after dosing
Radioactivity in whole blood and in plasma: AUC from time of dosing to the last quantifiable concentration (AUClast) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 312, 360, 408, 456, and 504 hours after radioactive dose. If subjects are not discharged on Day 22, blood will be collected at 576 and 648 hours after dosing
Radioactivity in whole blood and in plasma: Maximum concentration (Cmax) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 312, 360, 408, 456, and 504 hours after radioactive dose. If subjects are not discharged on Day 22, blood will be collected at 576 and 648 hours after dosing
Radioactivity in whole blood and in plasma: Time to Attain Cmax (tmax) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 312, 360, 408, 456, and 504 hours after radioactive dose. If subjects are not discharged on Day 22, blood will be collected at 576 and 648 hours after dosing
Radioactivity in whole blood and in plasma: Apparent terminal elimination half-life (t1/2) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 312, 360, 408, 456, and 504 hours after radioactive dose. If subjects are not discharged on Day 22, blood will be collected at 576 and 648 hours after dosing
Radioactivity in emesis (if applicable) | After study drug administration Days 1 up through 29
Radioactivity ratio blood/plasma | Day 1
Excretion ratio and cumulative excretion of radioactivity in urine | Pre-dose and after dosing collection times: 0 to 6, 6 to 12, 12 to 24, and in 24 hour intervals up to 504 hours after radioactive dose. If subjects are not discharged on Day 22, sample collection will continue in 24 hour intervals until discharge
Excretion ratio and cumulative excretion of radioactivity in feces | Pre-dose and after dosing in 24 hour intervals up to 504 hours after radioactive dose. If subjects are not discharged on Day 22, sample collection will continue in 24 hour intervals until the day of discharge

SECONDARY OUTCOMES:
Pharmacokinetic profile of isavuconazole in plasma: AUCinf, AUClast, Cmax, tmax, Apparent body clearance after dosing (CL/F), Apparent volume of distribution (Vz/F), t1/2 | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 312, 360, 408, 456, and 504 hours after radioactive dose. If subjects are not discharged on Day 22, blood will be collected at 576 and 648 hours after dosing
Pharmacokinetic Profile of isavuconazole in urine: Ae, Ae%, CLR | Pre-dose and 0 to 6, 6 to 12, 12 to 24, in 24 hour intervals up to 504 hours after radioactive dose. If subjects are not discharged on Day 22, sample collection will continue in 24 hour intervals until day of discharge
  Amount excreted (Ae), Percent of unchanged drug excreted into the urine (Ae%), Renal clearance (CLR)
Metabolic profile of isavuconazole and possible metabolites in plasma, urine, and feces | 8, 24,72, 144, and 312 hours after dosing. If subjects are not discharged on Day 22, samples will be taken at 504 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Covance, Madison, Wisconsin, United States